CLINICAL TRIAL: NCT04342988
Title: Effect of Cequa Treatment on Accuracy of Pre-operative Biometry and Higher Order Aberrations in Dry Eye Patients Undergoing Cataract Surgery
Brief Title: Effect of Cequa Treatment on Accuracy of Pre-operative Biometry & Higher Order Aberrations in Dry Eye Patients Undergoing Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Research Insight LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sun Cequa Accuracy 191118
Record Dates: First submitted 2020-04-06; First posted 2020-04-13 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2020-04

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cequa Treatment In Cataract Patients with Dry Eye Disease (Other): Duration of Study Treatment - 4 weeks All patients will receive cyclosporine ophthalmic solution (0.09%) BID in both eyes for 28 days, 1 drop per dose. Dosing will be BID, both eyes, assuming both eyes will eventually undergo cataract surgery. Otherwise, single eye treatment in the operative eye will be permitted.
  Interventions: Drug: Cequa

INTERVENTIONS:
Drug: Cequa — The effect of Cequa treatment on the accuracy of pre-operative biometry and on corneal higher-order aberrations (HOAs) in cataract patients who have signs of dry eye disease.

SUMMARY:
The purpose of this study is to examine the effect of Cequa treatment on the accuracy of pre-operative biometry and on corneal higher-order aberrations (HOAs) in cataract patients who have signs of dry eye disease.

DETAILED DESCRIPTION:
Hypothesis: In patients with dry eye, defined as corneal staining and a reduced tear breakup time, the accuracy of pre-operative biometry and corneal surface HOAs will improve significantly after four weeks of Cequa treatment.

Primary Outcome Measure: Spherical equivalent prediction error of pre-Cequa vs post-Cequa ocular biometry performed for cataract surgery.

Secondary Outcome Measures:

The impact of Cequa treatment on corneal higher order aberrations measured in the central 6 mm of the cornea.

The difference in SPEED questionnaire scores before and 4 weeks after Cequa treatment.

The difference in corneal staining and tear breakup time (TBUT) before and after treatment with Cequa.

ELIGIBILITY:
Inclusion Criteria:

* Patients with planned cataract surgery,
* The presence of central or inferior corneal fluorescein staining defined by the Oxford Scale
* Reduced tear break up time (TBUT) ≤ 10 seconds.
* Able to comprehend and sign a statement of informed consent.
* Willing and able to complete all required postoperative visits.

Exclusion Criteria:

* Ocular surgery (e.g., intraocular, oculoplastic, corneal or refractive surgical procedure) performed within the last 3 months or at any time that in the investigator's clinical judgment if it would interfere with the outcome measures of this study.
* Clinically significant ocular trauma.
* Active ocular Herpes simplex or Herpes Zoster infection
* Ocular inflammation (uveitis, iritis, scleritis, episcleritis, keratitis, conjunctivitis) at the discretion of the investigator.
* Ocular infection (e.g., viral, bacterial, mycobacterial, protozoan or fungal infection or the cornea, conjunctiva, lacrimal gland, lacrimal sac or eyelids including hordeolum/stye).
* Active, systemic or local disease condition that causes clinically significant ocular surface irritation such that it could interfere with the study findings.
* Moderate to severe (Grade 2-4) allergic, vernal or giant papillary conjunctivitis.
* Severe (Grade 3 or 4) inflammation of the eyelid (e.g., blepharochalasis, staphylococcal blepharitis or seborrheic blepharitis)
* Eyelid abnormalities that significantly affect the lid function (e.g., entropion, ectropion, tumor, edema, blepharospasm, lagophthalmos, severe trichiasis, severe ptosis).
* Ocular surface abnormality that may compromise the corneal integrity (e.g., prior chemical burn, recurrent corneal erosion, corneal epithelial defect, Grade 3 corneal fluorescein staining, map dot fingerprint dystrophy, or the effect of any other ophthalmic medication that might in the opinion of the investigator compromise the ocular surface integrity).
* Participation in this trial in the same patient's fellow eye
* Patients who are under age 18, pregnant or breastfeeding, or who may become pregnant during participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Spherical equivalent prediction error of pre-Cequa vs post-Cequa ocular biometry performed for cataract surgery. | Four weeks

SECONDARY OUTCOMES:
The impact of Cequa treatment on corneal higher order aberrations measured in the central 6 mm of the cornea. | Four Weeks
The difference in SPEED questionnaire scores before and 4 weeks after Cequa treatment. | Four Weeks
  To compare the difference in Standard Patient of Eye Dryness Questionnaire (SPEED) scores before and after 4 weeks of therapy with Cequa BID among patients with significant dry eye (decreased TBUT or corneal staining) with planned cataract surgery. The SPEED questionnaire gives a score from 0-28 that is the result of 8 items that assess frequency and severity of symptoms. Speed Score Severity rating: 0-4 Mild, 5-7 Moderate, 8+ Severe.
The difference in corneal staining before and after treatment with Cequa. | Four Weeks
  The presence of central or inferior corneal fluorescein staining defined by the Oxford Scale.
The difference in tear breakup time (TBUT) before and after treatment with Cequa. | Four Weeks
  Reduced tear break up time (TBUT) ≤ 10 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: John Hovanesian, MD, Study Director — Research Insight LLC
Locations (3):
- United States (3):
  - Harvard Eye Associates, Laguna Hills, California
  - Ophthalmology Associates, St Louis, Missouri
  - Ophthalmic Surgeons & Consultants of Ohio, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with, the Sponsor, and such that confidential or proprietary information is not disclosed

REFERENCES:
- [Background] Behrens A, Doyle JJ, Stern L, Chuck RS, McDonnell PJ, Azar DT, Dua HS, Hom M, Karpecki PM, Laibson PR, Lemp MA, Meisler DM, Del Castillo JM, O'Brien TP, Pflugfelder SC, Rolando M, Schein OD, Seitz B, Tseng SC, van Setten G, Wilson SE, Yiu SC; Dysfunctional tear syndrome study group. Dysfunctional tear syndrome: a Delphi approach to treatment recommendations. Cornea. 2006 Sep;25(8):900-7. doi: 10.1097/01.ico.0000214802.40313.fa. PMID 17102664
- [Background] Geerling G, Tauber J, Baudouin C, Goto E, Matsumoto Y, O'Brien T, Rolando M, Tsubota K, Nichols KK. The international workshop on meibomian gland dysfunction: report of the subcommittee on management and treatment of meibomian gland dysfunction. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):2050-64. doi: 10.1167/iovs.10-6997g. No abstract available. PMID 21450919